CLINICAL TRIAL: NCT01408719
Title: Effect of Beta-Glucan Molecular Weight and Viscosity on the Mechanism of Cholesterol Lowering in Humans
Brief Title: Effect of Beta-Glucan on Cholesterol Lowering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Nancy Ames, Research Scientist & Adjunct Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B2010:216
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Hypercholesterolemia
Keywords: Beta-Glucan; Barley; Molecular Weight; Viscosity; Cholesterol; Stable isotope; Gene-nutrient interaction; Gut microbiota
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5g LMW beta glucan (Experimental): 5 gram low molecular weight barley beta-glucan diet for 35 days
  Interventions: Dietary Supplement: Control
- 3g HMW beta glucan (Experimental): 3 gram high molecular weight barley beta-glucan diet for 35 days
  Interventions: Dietary Supplement: 3g LMW beta-glucan
- 3g LMW beta glucan (Experimental): 3 grams of low molecular weight beta-glucan diet for 35 days
  Interventions: Dietary Supplement: 5g LMW beta-glucan
- Control (Placebo Comparator): control diet containing negligible amount of beta glucan
  Interventions: Dietary Supplement: 3g HMW beta-glucan

INTERVENTIONS:
Dietary Supplement: Control — Minimal beta-glucan
  Arms: 5g LMW beta glucan
Dietary Supplement: 3g LMW beta-glucan — 3grams beta-glucan
  Arms: 3g HMW beta glucan
Dietary Supplement: 5g LMW beta-glucan — 5 grams beta-glucan
  Arms: 3g LMW beta glucan
Dietary Supplement: 3g HMW beta-glucan — 3 grams of high molecular weight beta-glucan
  Arms: Control

SUMMARY:
The primary aim of this study is to determine whether the cholesterol-lowering efficacy of barley b- glucan varied as function of molecular weight (MW) and the total daily amount consumed. Our second aim is to investigate the mechanism responsible for the action, specifically, whether β-glucan lowers circulating cholesterol concentration via inhibiting cholesterol absorption and synthesis. Thirdly, we aim to determine if any gene-diet interactions are associated with cholesterol lowering by barley β-glucan. In addition, we aim to investigate the alteration of the gut microbiota after β-glucan consumption and the correlation between the altered gut microbiota and cardiovascular disease risk factors.

DETAILED DESCRIPTION:
This study consists of four dietary phases which are separated by >28 days wash-out period. During the treatment phase, participants will be provided with all meals for the 35 day period. Breakfast meals will be consumed under the supervision of the research staff and lunch, dinner and snacks will be provided to take home in take-out packaging. While subjects are on the wash-out period they will return to their normal diet. The meals are on a 7 day rotating schedule that reflect an average Canadian diet. Changes in blood lipids, body weight, and waist circumference will be measured during each treatment phase. Cholesterol absorption and synthesis will be examined by stable isotope method. Single nucleotide polymorphisms (SNPs), rs3808607 of gene CYP7A1and rs429358 and rs7412 will be determined byTaqMan® SNP Genotyping assay following the manufacturer's protocol. Fecal samples will be collected at the end of each intervention phase and will be subjected to Illumina sequencing of 16S rRNA genes.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-40 kg/m2
* Fasting cholesterol levels of 5.0-8.0 mmol/L
* Fasting serum LDL cholesterol levels of 2.7-5.0 mmol/L

Exclusion Criteria:

* Pregnant or lactating
* Taking lipid lowering medication or nutritional supplements that affect blood lipids
* Dietary restrictions which would affect consuming the study diet for 5-wk for four study phases.
* Not deemed healthy by study physician

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, PhD, Principal Investigator — AAFC
Locations (1):
- Richardson Centre for Functional Foods and Neutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Wang Y, Harding SV, Eck P, Thandapilly SJ, Gamel TH, Abdel-Aal el-SM, Crow GH, Tosh SM, Jones PJ, Ames NP. High-Molecular-Weight beta-Glucan Decreases Serum Cholesterol Differentially Based on the CYP7A1 rs3808607 Polymorphism in Mildly Hypercholesterolemic Adults. J Nutr. 2016 Apr;146(4):720-7. doi: 10.3945/jn.115.223206. Epub 2016 Mar 2. PMID 26936139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Richardson Centre for Functionals Foods and Nutraceuticals, University of Manitoba, Winnipeg during July 2010 to May 2011
Pre-assignment Details: Over 200 subjects were screened; 45 subjects were enrolled in the study and randomly assigned to the experimental diets (treatment groups).
Groups:
- Sequence 1: 3g LMW followed by control, followed by 3g HMW, followed by 5g LMW
- Sequence 2: Control, followed by 3g HMW, followed by 5g LMW, followed by 3g LMW
- Sequence 3: 3g LMW, followed by 3g HMW, followed by 5g LMW, followed by control
- Sequence 4: 5g LMW, followed by 3g LMW, followed by 3g HMW, followed by control
- Sequence 5: 3g HMW, followed by 3g LMW, followed by control, followed by 5g LMW
- Sequence 6: control, followed by 5g LMW, followed by 3g HMW, followed by 3g LMW
- Sequence 7: 5g LMW, followed by 3g LMW, followed control, followed by 3g HMW
- Sequence 8: 3g LMW, followed by 3g HMW, followed by control, followed by 5g HMW
- Sequence 9: Control, followed by 5g HMW, followed by 3g LMW, followed by 3g HMW
- Sequence 10: Control, followed by 3g LMW, followed by 5g LMW, followed by 3g HMW
- Sequence 11: 3g HMW, followed by control, followed by 5g LMW, followed by 3g LMW
- Sequence 12: 5g LMW, followed by control, followed by 3g LMW, followed by 3g HMW
- Sequence 13: 3g HMW, followed by control, followed by 3g LMW, followed by 5g LMW
- Sequence 14: 3g LMW, followed by 5g LMW, followed by 3g HMW, followed by control
- Sequence 15: 3g LMW, followed by 5g LMW, followed by control, followed by 3g HMW
- Sequence 16: 3g HMW, followed by 5g LMW, followed 3g LMW, followed by control
- Sequence 17: 3g HMW, followed by 3g LMW, followed 5g LMW, followed by control
- Sequence 18: 5g LMW, followed by 3g HMW, followed by control, followed by 3g LMW
- Sequence 19: Control, followed by 3g HMW, followed by 3g LMW, followed by 5g LMW
- Sequence 20: 3g HMW, followed by 5g LMW, followed by control, followed by 3g LMW
Period: First Intervention (35 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 2 | 2 | 4 | 3 | 2 | 3 | 2 | 1 | 2 | 2 | 2 | 5 | 1 | 2 | 3 | 2 | 1 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 2 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Period: Washout Period (28 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 2 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 2 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (35 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 2 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 2 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (28 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (35 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (28 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention (35 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Completed | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: It is a cross over trial so the total number of participants is same throughout the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20 | Total
Number analyzed (Participants) | 2 | 3 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 1 | 1 | 1 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15.6) | 52.7 (3.5) | 40 (0) | 63 (1.4) | 70 (10.6) | 55 (14) | 55.5 (2.12) | 67 (1.4) | 57 (0) | 27 (0) | 62.5 (0.7) | 59.5 (4.9) | 62 (0) | 59.3 (3.8) | 76 (0) | 58 (0) | 53 (8.5) | 59 (0) | 65 (0) | 59 (0) | 57.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 20
  Male | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Changs in Total Cholesterol
Description: Fasted total cholesterol concentration will be measured using the automated enzymatic methods.
Time Frame: Beginning and end of each phase
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | 5g LMW Beta Glucan | 3g HMW Beta Glucan | 3g LMW Beta Glucan | Control
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmol/L | -0.42 (0.09) | -0.60 (0.09) | -0.46 (0.09) | -0.30 (0.09)

2. Secondary Outcome: Cholesterol Absorption/Synthesis
Description: The rate of cholesterol absorption and synthesis will be measured in each intervention phase using single stable isotope labelling technique.
Time Frame: End of each phase
Reporting Status: Not Posted

3. Secondary Outcome: Potential Gene-nutrient Interactions: CYP7A1 and APOE
Description: The Single Nucleotide Polymorphism (SNP) rs3808607 of CYP7A1 gene, rs429358 and rs7412 of APOE gene, and their associations with different blood lipid responses to beta-glucan interventions will be determined.
Time Frame: Once for each participant
Reporting Status: Not Posted

4. Primary Outcome: Changes in LDL Cholesterol
Description: Serum LDL cholesterol will be estimated using the Friedewald equation.
Time Frame: Beginning and end of each phase
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Body Weight and Waist Circumference(WC)
Description: Body weight will be monitored every day when subject visits the Richardson Centre. Waist circumference will be measured at the beginning and end of each study phase.
Time Frame: Every day for body weight; beginning and end of each phase for WC
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Control: Minimal barley and minimal beta-glucan
- 3g HMW Beta-glucan: 3 grams high molecular weight barley beta-glucan
- 3g LMW Beta-glucan: 3 grams low molecular weight barley beta-glucan
- 5g LMW Beta-glucan: 5 grams low molecular weight barley beta-glucan
Arm/Group | Control | 3g HMW Beta-glucan | 3g LMW Beta-glucan | 5g LMW Beta-glucan
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes